CLINICAL TRIAL: NCT07009626
Title: Effectiveness of Simulation in Shoulder Dystocia Management Education: A Randomized-Controlled Trial
Brief Title: Simulation in Shoulder Dystocia Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, yasemin hamlacı başkaya, Assoc. prof., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 28052025
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Dystocia; Simulation Based Medical Education; Midwifery
Keywords: shoulder dystocia; simulation; midwifery education; anxiety
MeSH Terms: conditions — Shoulder Dystocia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group: The instructor will position the pelvic mannequin so that the fetus is in vertex presentation. A person independent of the research and training will facilitate the descent of the baby into the pelvic mannequin. After the delivery of the baby's head, the baby's descent will be stopped and the instructor will not allow the baby to be born. Each student will be given the opportunity to practice the process on the mannequin according to the steps of shoulder dystocia management. Each practice session will last approximately 10 minutes. The researcher will observe each student and provide feedback on their performance, including discussion of any errors made.
- Computer-based high-validity birth simulator group (Experimental): Computer-based high-validity birth simulator group: The instructor will place the fetus in a computer-based full-body birthing manikin in vertex presentation. In addition, the pregnant woman will be vocalized to increase realism and the patient's vital signs, fetal heart rate, etc. will be displayed on the patient monitor. The same scenario will be initiated for each student in the simulation group. Each student will be given the opportunity to practice the process on the simulation model in accordance with the shoulder dystocia delivery management steps. Each practice session will last 15-20 minutes. The researcher will observe each student and provide feedback on their performance, including discussion of any errors made.
  Interventions: Other: Computer-based high-validity birth simulator

INTERVENTIONS:
Other: Computer-based high-validity birth simulator — Computer-based high-validity birth simulator: All students in the intervention group underwent the same scenario of birth. Initially, the aim was to diagnose shoulder dystocia by ensuring that the shoulders were not delivered after the fetal head was delivered.
  Arms: Computer-based high-validity birth simulator group

SUMMARY:
Shoulder dystocia is an unpredictable and unpredictable emergency obstetric condition that causes serious maternal and neonatal complications. Therefore, it requires immediate and effective intervention. It is known as the condition in which the shoulders cannot be released from the pelvis and remain stuck after the fetal head is born during delivery. Fetal macrosomia is shown as the most important risk factor for shoulder dystocia. The intervention to be performed for shoulder dystocia should start from the least invasive and progress to the more invasive. Detection and management of shoulder dystocia requires sufficient technical knowledge, skills and experience. Simulation-based learning in midwifery education and practice provides students with the opportunity to manage and develop skills in many risky situations close to reality outside the hospital environment. In addition, the fact that the application can be repeated many times without harming people also affects the anxiety and self-efficacy levels of students before real clinical experience. As a result, it is understood that shoulder dystocia is an important condition that cannot be predicted and prevented, has very serious maternal and neonatal consequences, and a systematic approach should be used in its prevention, early diagnosis and management. The aim of this study is to evaluate the effect of a computer-based simulation training model on the knowledge level, management skills and anxiety levels of midwifery students about shoulder dystocia. The study will be conducted with all students enrolled in the "Risky Birth and Postpartum Period" course at the Department of Midwifery, Faculty of Health Sciences, Sakarya University in the 2024-2025 academic year. Data in the study will be collected through the Student Identification Form, Shoulder Dystocia and Management Information Form, Shoulder Dystocia Management Individual Assessment Form and Shoulder Dystocia Management Skills Assessment Form. The analysis of the data obtained from the study will be done with the SPSS program. It is thought that the study will make a significant contribution to the literature in terms of evaluating the effect of the computer-based simulation training model on shoulder dystocia management.

DETAILED DESCRIPTION:
Shoulder dystocia is defined as failure to deliver the shoulders after the delivery of the fetal head. This condition may occur as a result of a mismatch between the fetal shoulder size and the pelvic inlet, and may develop as an anterior or posterior shoulder attachment, or it may be seen in both shoulders. This condition is an unpredictable and unavoidable obstetric emergency, occurring in 0.6% to 1.4% of births. Shoulder dystocia usually includes risk factors such as maternal obesity, fetal macrosomia, maternal diabetes, prolonged labor, advanced age, use of epidural anesthesia, and a history of dystocia in previous births. Transient brachial plexus injury (BPI) is the most common fetal complication due to shoulder dystocia. Other fetal complications include clavicle and humerus injuries, permanent BPI, hypoxic ischemic encephalopathy and death. Maternal complications can lead to vaginal and cervical lacerations, postpartum hemorrhage, II.-III.-IV. degree perineal tears, and even late-term fistulas. Therefore, it is vital to know the risk factors in advance and to ensure the order of maneuvers to be performed and the correct application skills for difficult births that occur. Simulation education has been used in the health field for many years. Simulators help with rapid critical thinking and management of situations that cause confusion. In skill-based midwifery education, simulation-based learning focuses on many risky situations such as postpartum hemorrhage, shoulder impingement, and emergency breech delivery. The use of computer-based simulators allows students to practice and develop their skills in an environment that is almost like a hospital before going to hospital practice. Computer-based simulators are quite educational for students because they provide opportunities for realistic errors and realistic error attempts. Simulators are also known to increase learning satisfaction, improve communication skills and increase self-efficacy. In this study, it was aimed to evaluate the effect of the computer-based simulation training model on the knowledge level, management skills and anxiety levels of midwifery students about shoulder dystocia.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the midwifery department,
* Attending the risky birth and postpartum period course,
* Agreeing to participate in the study

Exclusion Criteria:

* Those who have previously taken the risky birth and postpartum period course and failed the course,
* Those who did not attend the shoulder dystocia management course,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Shoulder Dystocia and Management Information Form | pre-intervention, 1 hour after intervention
  This is a questionnaire form developed by researchers in line with the information in the guide developed by RCOG for the management of shoulder dystocia. This form, which will be applied before and after the training, consists of 18 questions. It was used to determine the knowledge levels of students about shoulder dystocia and its management. One point was given for each correct answer given to the questions in the survey. The maximum total score that can be obtained is 18. Students will mark the questions in the shoulder dystocia and its management information form as true, false or I have no idea.
State Anxiety Inventory | pre-intervention, 1 hour after intervention
  The inventory developed by Spielberger and colleagues (1970) is a self-assessment questionnaire consisting of short assessments (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). The validity and reliability of the inventory in Turkey was conducted by Öner and Lecompte (1983) (Öner & Le Compte, 1983). The State Anxiety Inventory consists of 20 items and requires the individual to answer how he/she feels at a certain moment and under certain conditions, taking into account his/her feelings about the situation he/she is in. The scale is a Likert-type scale with four points ranging from "Not at all" to "Completely". High scores indicate a high level of anxiety, and low scores indicate a low level of anxiety. In the validity and reliability study of the inventory, the Cronbach Alpha coefficient for the SAI was between 0.94 and 0.96 (Öner & Le Compte, 1983).
Shoulder Dystocia Management Skills Assessment Form | 1 hours
  It is a form that evaluates students' implementation of the steps in shoulder dystocia management.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Hamlacı Başkaya, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grobman WA. Shoulder dystocia: simulation and a team-centered protocol. Semin Perinatol. 2014 Jun;38(4):205-9. doi: 10.1053/j.semperi.2014.04.006. PMID 24863026
- [Background] Gurewitsch Allen ED. Simulation of Shoulder Dystocia for Skill Acquisition and Competency Assessment: A Systematic Review and Gap Analysis. Simul Healthc. 2018 Aug;13(4):268-283. doi: 10.1097/SIH.0000000000000292. PMID 29381590
- [Background] Hill DA, Lense J, Roepcke F. Shoulder Dystocia: Managing an Obstetric Emergency. Am Fam Physician. 2020 Jul 15;102(2):84-90. PMID 32667171
- [Background] Hill MG, Cohen WR. Shoulder dystocia: prediction and management. Womens Health (Lond). 2016;12(2):251-61. doi: 10.2217/whe.15.103. Epub 2016 Feb 22. PMID 26901875
- [Background] Behram, M., ve Eyi, EGY. Vajinal Doğum Sırasında Omuz Distosisi Gelişen Olguların Değerlendirilmesi. Internatıonal Anatolıa Academıc Onlıne Journal, Health Scıences, 2021; 7(2), 109-118.
- [Background] Nassar AK, Al-Manaseer F, Knowlton LM, Tuma F. Virtual reality (VR) as a simulation modality for technical skills acquisition. Ann Med Surg (Lond). 2021 Oct 27;71:102945. doi: 10.1016/j.amsu.2021.102945. eCollection 2021 Nov. PMID 34840738
- [Background] Padilha JM, Machado PP, Ribeiro A, Ramos J, Costa P. Clinical Virtual Simulation in Nursing Education: Randomized Controlled Trial. J Med Internet Res. 2019 Mar 18;21(3):e11529. doi: 10.2196/11529. PMID 30882355
- [Background] Şenoğlu, A., ve Karaçam, Z. Omuz Distosisi: Ebelik Eğitim ve Uygulamalarındaki Yeri. Lokman Hekim Dergisi, 2019;9 (2): 147-159 DOI: 10.31020/mutftd.522365